CLINICAL TRIAL: NCT00975676
Title: A Substudy of the IBCSG 24-02/ SOFT Trial to Investigate Estrogen Suppression for Patients Participating in Arms B and C of the IBCSG 24-02/ SOFT Trial
Brief Title: Study of Estrogen Levels in Premenopausal Women Who Have Undergone Surgery for Breast Cancer and Are Receiving Triptorelin and Tamoxifen Citrate or Exemestane on Clinical Trial IBCSG 24-02
Acronym: SOFT-EST
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: ETOP IBCSG Partners Foundation (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000650841; IBCSG 24-02-SOFT-EST; SOLTI 0801; BIG 2-02
Record Dates: First submitted 2009-09-10; First posted 2009-09-11 (Estimated); Results first posted 2021-10-25 (Actual); Last update posted 2021-10-25 (Actual); Status verified 2021-09

CONDITIONS: Breast Cancer
Keywords: estrogen receptor-positive breast cancer; progesterone receptor-positive breast cancer; stage IA breast cancer; stage IB breast cancer; stage II breast cancer; stage IIIA breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Chromatography, Gas

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Triptorelin plus tamoxifen (Experimental): Determination of estrogen levels in blood samples from patients being treated with triptorelin plus tamoxifen for 5 years.
  Interventions: Other: gas chromatography / tandem mass spectometry
- Triptorelin plus exemestane (Experimental): Determination of estrogen levels in blood samples from patients being treated with triptorelin plus exemestane for 5 years.
  Interventions: Other: gas chromatography / tandem mass spectometry

INTERVENTIONS:
Other: gas chromatography / tandem mass spectometry — Determination of estrogen levels through gas chromatography.

SUMMARY:
RATIONALE: Studying samples of blood from patients with breast cancer in the laboratory may help doctors learn how well triptorelin given together with tamoxifen citrate or exemestane works in lowering estrogen levels.

PURPOSE: This clinical trial is studying estrogen levels in premenopausal women who have undergone surgery for breast cancer and are receiving triptorelin and tamoxifen citrate or exemestane on clinical trial IBCSG-2402.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Describe estrogen levels (estradiol [E2], estrone [E1], and estrone sulphate [E1S]) at different time points during the first 4 years of treatment with triptorelin in combination with either tamoxifen citrate or exemestane on clinical trial IBCSG-2402 in premenopausal women with resected breast cancer.
* Assess whether there is a suboptimally estrogen-suppressed subgroup of patients who receive exemestane.

Secondary

* Compare estrogen levels (E2, E1, E1S) at different time points during treatment with triptorelin in combination with either tamoxifen citrate or exemestane.
* Examine potential predictive factors of ineffective estrogen suppression (e.g., age, chemotherapy [yes/no], type of chemotherapy received, smoking history, BMI, and evidence of menses at study entry).
* Investigate the predictive value of optimal estrogen suppression during the first 6 and 12 months of treatment with regard to long-term estrogen suppression (4-year period).
* Compare disease-free survival of suboptimally estrogen-suppressed patients treated with exemestane with that of patients with optimal suppression (exploratory analysis).
* Examine related endocrine function (FSH and LH) to further elucidate causes of suboptimal estrogen suppression.

OUTLINE: This is a multicenter study.

Blood samples are collected at baseline and at 3, 6, 12, 18, 24, 36, and 48 months for measurement of estrogen levels (estradiol [E2], estrone [E1], and estrone sulphate [E1S]) by gas chromatography-mass spectrometry and measurement of endocrine function (FSH and LH).

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed resected breast cancer
* Concurrent enrollment on clinical trial IBCSG-2402 (SOFT trial) required

  * Randomized to receive triptorelin in combination with either tamoxifen citrate or exemestane
* Hormone receptor status:

  * Estrogen receptor- and/or progesterone receptor-positive tumor

PATIENT CHARACTERISTICS:

* Premenopausal

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics

Ages: 0 Years to 120 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 123 (Actual)
Dates: Start 2008-11-25; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Prudence Francis, MD, Study Chair — Peter MacCallum Cancer Centre, Australia
Locations (24):
- Centre Rene Huguenin, Saint-Cloud, France
- National Institute of Oncology, Budapest, Hungary
- Italy (2):
  - Salvatore Maugeri Foundation, Pavia
  - Clinica Oncologica, Policlinico Univeritario, Udine
- INEN (Instituto de Enfermedades Neoplasicas), Lima, Peru
- Centro de Lisboa, Lisbon, Portugal
- Spain (13):
  - Vall d'Hebron University Hospital, Barcelona
  - Hospital Clinic i Provincial de Barcelona, Barcelona
  - Hospital Dr Negrin, Las Palmas de Gran Canaria
  - H.U. Arnau de Vilanova, Lleida
  - Centro Oncologico Md Anderson, Madrid
  - Hospital Ramon Y Cajal, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Son Dureta, Palma
  - Hospital Son Llatzer, Palma
  - Hospital Sant Joan de Reus, Reus
  - Hospital Sant Pau i Santa Tecla, Tarragona
  - Hospital Clinico Universitario de Valencia, Valencia
  - Instituto Valenciano de Oncologia, Valencia
- Sahlgrenska University Hospital Gothenburg, Gothenburg, Sweden
- Switzerland (4):
  - Kantonsspital Graubünden, Chur
  - Multidisciplinary Oncology Centre, CHUV, Lausanne
  - Spital Thun, Thun
  - Brust-Zentrum, Zurich

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The SOFT-EST substudy was activated on 25 Nov 2008. Participating Centers were expected to enroll all or most patients who planned to use triptorelin as method of OFS, if randomized to receive OFS, into this substudy. The accrual goal for the substudy was 120 patients (30 T+OFS; 90 E+OFS). Enrollment of 30 patients randomly assigned to T+OFS was reached by 31 Dec 2009; enrollment of patients randomly assigned to E+OFS continued until SOFT and SOFT-EST enrollment closed on 31 Jan 2011.
Groups:
- Triptorelin Plus Tamoxifen: Determination of estrogen levels in blood samples from patients being treated with triptorelin plus tamoxifen for 5 years. The final analytic cohort included 109 patients from the intent to treat (ITT) population, who had ≥2 samples assayed or E+Trip=83, T+Trip=26 respectively, patients with only baseline data were excluded.
- Triptorelin Plus Exemestane: Determination of estrogen levels in blood samples from patients being treated with triptorelin plus exemestane for 5 years. The final analytic cohort included 109 patients from the intent to treat (ITT) population, who had ≥2 samples assayed or E+Trip=83, T+Trip=26 respectively, patients with only baseline data were excluded.
Period: Overall Study
Arm/Group | Triptorelin Plus Tamoxifen | Triptorelin Plus Exemestane
Started | 32 | 91
Completed | 26 | 83
Not Completed | 6 | 8
Not completed — Baseline samples only, no sample analyzed or only single sample available | 6 | 8

BASELINE CHARACTERISTICS:
Population: Intent to treat (ITT) population: all patients receiving triptorelin plus either tamoxifen (T+Trip) or exemestane (E+Trip) with the exception of patients who withdrew consent and/or never started triptorelin. Analysis cohort (N=109): all patients from ITT population, who had two sample data were included, given the primary aims of this analysis is for the long term (4 years) data, patients with only baseline data were excluded. Fourteen patients were excluded.
Groups:
- Total: Total of all reporting groups
Arm/Group | Triptorelin Plus Tamoxifen | Triptorelin Plus Exemestane | Total
Number analyzed (Participants) | 26 | 83 | 109
Age, Customized [Count of Participants; unit: Participants] — Population: Patient characteristics for the analytic cohort of 109 patients according to treatment assignment.
  Participants
    <35 | 0 | 8 | 8
    35-39 | 5 | 10 | 15
    40-44 | 7 | 26 | 33
    45-49 | 14 | 39 | 53
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26 | 83 | 109
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 25 | 81 | 106
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 2 | 3
Estradiol (E2), pg/mL [Mean (Standard Deviation); unit: pg/mL] — Population: Excludes 2 patients without baseline samples
  pg/mL
    number analyzed (Participants) | 26 | 81 | 107
    (all) | 109.81 (119.81) | 96.55 (151.23) | 99.78 (143.68)
Estrone (E1), pg/mL [Mean (Standard Deviation); unit: pg/mL] — Population: Excludes 2 patients without baseline samples
  pg/mL
    number analyzed (Participants) | 26 | 81 | 107
    (all) | 60.27 (52.40) | 65.42 (78.12) | 64.17 (72.52)
Estrone sulfate (E1S), pg/mL [Mean (Standard Deviation); unit: pg/mL] — Population: Excludes 2 patients without baseline samples
  pg/mL
    number analyzed (Participants) | 26 | 81 | 107
    (all) | 1437.02 (1825.06) | 1371.21 (1763.84) | 1387.20 (1770.42)
Follicle-stimulating hormone (FSH), LU/L [Mean (Standard Deviation); unit: LU/L] — Population: Excludes 6 patients without baseline samples
  LU/L
    number analyzed (Participants) | 25 | 78 | 103
    (all) | 25.14 (29.05) | 30.30 (27.37) | 29.05 (27.73)
Luteinizing hormone (LH), LU/L [Mean (Standard Deviation); unit: LU/L] — Population: Excludes 5 patients without baseline samples
  LU/L
    number analyzed (Participants) | 25 | 79 | 104
    (all) | 16.77 (16.29) | 18.97 (16.12) | 18.44 (16.11)

OUTCOME MEASURES:

1. Primary Outcome: Estrogen Levels (Estradiol [E2], Estrone [E1], and Estrone Sulphate [E1S]) at Different Time Points During the First 4 Years of Treatment With Triptorelin (Trip) in Combination With Either Tamoxifen (T) or Exemestane (E), IBCSG 24-02 SOFT-EST Substudy
Description: Estrogen levels (estradiol [E2], estrone [E1], and estrone sulphate [E1S]) were measured at the following time points for the SOFT-EST: 0 (baseline), 3, 6, 12, 18, 24, 36, and 48 months after randomization. Some of these samples were not used, including un-scheduled sample, post surgery or vaginal bleeding, samples taken post early discontinuation (ED) or discontinuation of GnRH injections.
Time Frame: 0 (baseline), 3, 6, 12, 18, 24, 36, and 48 months after randomization
Population: The final (4 years) analysis cohort (N=109) consists of all patients from the intent to treat (ITT) population (N=123) who had at least 2 samples analyzed and who received at least one GnRH analogue triptorelin injection during follow-up. Fourteen patients were excluded due to the reasons of 1) never start TE and never received GnRH (gonadotropin-releasing hormone) analogue triptorelin; 2) only baseline sample available; 3) single sample at 24 months; 4) patients without sample analyzed.
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Triptorelin Plus Tamoxifen | Triptorelin Plus Exemestane
Number analyzed (Participants) | 26 | 83
pg/mL
  Estradiol (E2) levels at baseline (0 months): number analyzed (Participants) | 26 | 81
  Estradiol (E2) levels at baseline (0 months) | 109.81 (119.151) | 96.55 (151.235)
  Estradiol (E2) levels at 3 months: number analyzed (Participants) | 25 | 67
  Estradiol (E2) levels at 3 months | 4.876 (7.123) | 3.973 (8.439)
  Estradiol (E2) levels at 6 months: number analyzed (Participants) | 24 | 66
  Estradiol (E2) levels at 6 months | 3.761 (2.02) | 3.672 (8.006)
  Estradiol (E2) levels at 12 months: number analyzed (Participants) | 20 | 68
  Estradiol (E2) levels at 12 months | 4.013 (2.765) | 2.486 (5)
  Estradiol (E2) levels at 18 months: number analyzed (Participants) | 20 | 65
  Estradiol (E2) levels at 18 months | 7.306 (16.325) | 2.527 (6.204)
  Estradiol (E2) levels at 24 months: number analyzed (Participants) | 15 | 62
  Estradiol (E2) levels at 24 months | 4.453 (3.347) | 2.52 (6.566)
  Estradiol (E2) levels at 36 months: number analyzed (Participants) | 14 | 60
  Estradiol (E2) levels at 36 months | 3.704 (2.138) | 1.654 (2.764)
  Estradiol (E2) levels at 48 months: number analyzed (Participants) | 14 | 50
  Estradiol (E2) levels at 48 months | 5.914 (8.959) | 9.073 (57.307)
  Estrone (E1) levels at baseline (0 months): number analyzed (Participants) | 26 | 81
  Estrone (E1) levels at baseline (0 months) | 60.27 (52.4) | 65.42 (78.12)
  Estrone (E1) levels at 3 months: number analyzed (Participants) | 25 | 67
  Estrone (E1) levels at 3 months | 17.8 (6.73) | 2.93 (3.33)
  Estrone (E1) levels at 6 months: number analyzed (Participants) | 24 | 66
  Estrone (E1) levels at 6 months | 18.66 (7.54) | 2.73 (3.12)
  Estrone (E1) levels at 12 months: number analyzed (Participants) | 21 | 68
  Estrone (E1) levels at 12 months | 19.05 (8.4) | 3.71 (6.35)
  Estrone (E1) levels at 18 months: number analyzed (Participants) | 20 | 65
  Estrone (E1) levels at 18 months | 18.64 (9.35) | 8.47 (33.42)
  Estrone (E1) levels at 24 months: number analyzed (Participants) | 15 | 62
  Estrone (E1) levels at 24 months | 18.96 (7.63) | 4.69 (9.16)
  Estrone (E1) levels at 36 months: number analyzed (Participants) | 14 | 60
  Estrone (E1) levels at 36 months | 19.49 (7.32) | 4.93 (9.16)
  Estrone (E1) levels at 48 months: number analyzed (Participants) | 14 | 50
  Estrone (E1) levels at 48 months | 19.14 (7.24) | 8.53 (35.07)
  Estrone sulfate (E1S) levels at baseline (0 months): number analyzed (Participants) | 26 | 81
  Estrone sulfate (E1S) levels at baseline (0 months) | 1437 (1825.06) | 1371 (1763.84)
  Estrone sulfate (E1S) levels at 3 months: number analyzed (Participants) | 25 | 67
  Estrone sulfate (E1S) levels at 3 months | 281.4 (183.44) | 56.02 (133.71)
  Estrone sulfate (E1S) levels at 6 months: number analyzed (Participants) | 24 | 66
  Estrone sulfate (E1S) levels at 6 months | 259 (167.23) | 54.7 (97.66)
  Estrone sulfate (E1S) levels at 12 months: number analyzed (Participants) | 21 | 68
  Estrone sulfate (E1S) levels at 12 months | 278.5 (236.38) | 47.31 (130.45)
  Estrone sulfate (E1S) levels at 18 months: number analyzed (Participants) | 20 | 64
  Estrone sulfate (E1S) levels at 18 months | 281.8 (160.6) | 63.52 (175.19)
  Estrone sulfate (E1S) levels at 24 months: number analyzed (Participants) | 14 | 59
  Estrone sulfate (E1S) levels at 24 months | 242.6 (96.75) | 73.56 (258.29)
  Estrone sulfate (E1S) levels at 36 months: number analyzed (Participants) | 14 | 60
  Estrone sulfate (E1S) levels at 36 months | 249.4 (113.27) | 53.27 (151.03)
  Estrone sulfate (E1S) levels at 48 months: number analyzed (Participants) | 13 | 46
  Estrone sulfate (E1S) levels at 48 months | 231.1 (93.46) | 112 (556.81)

2. Primary Outcome: Number of Patients Who Receive Exemestane Experiencing Suboptimal Estrogen Suppression
Description: Suboptimal estrogen suppression (SES), estradiol (E2) levels greater than 2.72 pg/mL in at least 2 post-baseline samples.
Time Frame: 0 (baseline), 3, 6, 12, 18, 24, 36, and 48 months after randomization
Population: Among patients randomly assigned to exemestane + triptorelin and included in the analysis cohort (N=83), the number of patients who experienced suboptimal suppression at each timepoint, with 95% exact binomial confidence intervals (CI), were reported. Two patients were excluded due to no baseline sample.
Measure: Count of Participants; unit: Participants
Arm/Group | Triptorelin Plus Exemestane
Number analyzed (Participants) | 83
Participants
  Patients with E2 > 2.72 pg/mL at baseline (0 months): number analyzed (Participants) | 81
  Patients with E2 > 2.72 pg/mL at baseline (0 months) | 74
  Patients with E2 > 2.72 pg/mL at 3 months: number analyzed (Participants) | 67
  Patients with E2 > 2.72 pg/mL at 3 months | 17
  Patients with E2 > 2.72 pg/mL at 6 months: number analyzed (Participants) | 66
  Patients with E2 > 2.72 pg/mL at 6 months | 16
  Patients with E2 > 2.72 pg/mL at 12 months: number analyzed (Participants) | 68
  Patients with E2 > 2.72 pg/mL at 12 months | 12
  Patients with E2 > 2.72 pg/mL at 18 months: number analyzed (Participants) | 65
  Patients with E2 > 2.72 pg/mL at 18 months | 12
  Patients with E2 > 2.72 pg/mL at 24 months: number analyzed (Participants) | 62
  Patients with E2 > 2.72 pg/mL at 24 months | 8
  Patients with E2 > 2.72 pg/mL at 36 months: number analyzed (Participants) | 60
  Patients with E2 > 2.72 pg/mL at 36 months | 8
  Patients with E2 > 2.72 pg/mL at 48 months: number analyzed (Participants) | 49
  Patients with E2 > 2.72 pg/mL at 48 months | 3

3. Secondary Outcome: Comparison of Estrogen Levels at Different Time Points During Treatment
Description: Percent (%) change of estrogen levels estradiol (E2), estrone (E1), and estrone sulphate (E1S) at each timepoint from baseline: e.g. {E2(t)-E2(0)} / E2(0)*100, where t= 3, 6, 12, 18, 24, 36, and 48 months from randomization
Time Frame: baseline (0 months), 3, 6, 12, 18, 24, 36, and 48 months from randomization
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percent change of estrogen levels
Arm/Group | Triptorelin Plus Tamoxifen | Triptorelin Plus Exemestane
Number analyzed (Participants) | 26 | 83
percent change of estrogen levels
  Percent change from baseline of estradiol (E2) at 0 months (baseline): number analyzed (Participants) | 26 | 81
  Percent change from baseline of estradiol (E2) at 0 months (baseline) | 0 (0) | 0 (0)
  Percent change from baseline of estradiol (E2) at 3 months: number analyzed (Participants) | 25 | 67
  Percent change from baseline of estradiol (E2) at 3 months | -70 (40) | -76 (75)
  Percent change from baseline of estradiol (E2) at 6 months: number analyzed (Participants) | 24 | 66
  Percent change from baseline of estradiol (E2) at 6 months | -69 (44) | -82 (62)
  Percent change from baseline of estradiol (E2) at 12 months: number analyzed (Participants) | 20 | 68
  Percent change from baseline of estradiol (E2) at 12 months | -57 (61) | -83 (47)
  Percent change from baseline of estradiol (E2) at 18 months: number analyzed (Participants) | 20 | 65
  Percent change from baseline of estradiol (E2) at 18 months | -61 (50) | -85 (37)
  Percent change from baseline of estradiol (E2) at 24 months: number analyzed (Participants) | 15 | 62
  Percent change from baseline of estradiol (E2) at 24 months | -63 (48) | -79 (61)
  Percent change from baseline of estradiol (E2) at 36 months: number analyzed (Participants) | 14 | 60
  Percent change from baseline of estradiol (E2) at 36 months | -56 (44) | -86 (33)
  Percent change from baseline of estradiol (E2) at 48 months: number analyzed (Participants) | 14 | 49
  Percent change from baseline of estradiol (E2) at 48 months | -65 (41) | -79 (87)
  Percent change from baseline of estrone (E1) at 0 months (baseline): number analyzed (Participants) | 26 | 81
  Percent change from baseline of estrone (E1) at 0 months (baseline) | 0 (0) | 0 (0)
  Percent change from baseline of estrone (E1) at 3 months: number analyzed (Participants) | 25 | 67
  Percent change from baseline of estrone (E1) at 3 months | -48 (41) | -90 (18)
  Percent change from baseline of estrone (E1) at 6 months: number analyzed (Participants) | 24 | 66
  Percent change from baseline of estrone (E1) at 6 months | -43 (50) | -90 (19)
  Percent change from baseline of estrone (E1) at 12 months: number analyzed (Participants) | 21 | 68
  Percent change from baseline of estrone (E1) at 12 months | -38 (55) | -81 (61)
  Percent change from baseline of estrone (E1) at 18 months: number analyzed (Participants) | 20 | 65
  Percent change from baseline of estrone (E1) at 18 months | -44 (37) | -75 (86)
  Percent change from baseline of estrone (E1) at 24 months: number analyzed (Participants) | 15 | 62
  Percent change from baseline of estrone (E1) at 24 months | -40 (43) | -84 (33)
  Percent change from baseline of estrone (E1) at 36 months: number analyzed (Participants) | 14 | 60
  Percent change from baseline of estrone (E1) at 36 months | -29 (39) | -82 (35)
  Percent change from baseline of estrone (E1) at 48 months: number analyzed (Participants) | 14 | 50
  Percent change from baseline of estrone (E1) at 48 months | -41 (33) | -70 (133)
  Percent change from baseline of estrone sulfate (E1S) at 0 months (baseline): number analyzed (Participants) | 26 | 81
  Percent change from baseline of estrone sulfate (E1S) at 0 months (baseline) | 0 (0) | 0 (0)
  Percent change from baseline of estrone sulfate (E1S) at 3 months: number analyzed (Participants) | 25 | 67
  Percent change from baseline of estrone sulfate (E1S) at 3 months | -43 (73) | -90 (27)
  Percent change from baseline of estrone sulfate (E1S) at 6 months: number analyzed (Participants) | 24 | 66
  Percent change from baseline of estrone sulfate (E1S) at 6 months | -50 (59) | -87 (35)
  Percent change from baseline of estrone sulfate (E1S) at 12 months: number analyzed (Participants) | 21 | 68
  Percent change from baseline of estrone sulfate (E1S) at 12 months | -35 (82) | -92 (17)
  Percent change from baseline of estrone sulfate (E1S) at 18 months: number analyzed (Participants) | 20 | 64
  Percent change from baseline of estrone sulfate (E1S) at 18 months | -35 (68) | -92 (16)
  Percent change from baseline of estrone sulfate (E1S) at 24 months: number analyzed (Participants) | 14 | 59
  Percent change from baseline of estrone sulfate (E1S) at 24 months | -27 (87) | -88 (33)
  Percent change from baseline of estrone sulfate (E1S) at 36 months: number analyzed (Participants) | 14 | 60
  Percent change from baseline of estrone sulfate (E1S) at 36 months | -26 (63) | -70 (173)
  Percent change from baseline of estrone sulfate (E1S) at 48 months: number analyzed (Participants) | 13 | 46
  Percent change from baseline of estrone sulfate (E1S) at 48 months | -36 (66) | -87 (53)

4. Secondary Outcome: Number of Participants With Potential Predictive Factors of Ineffective Estrogen Suppression
Description: Potential predictive factors of ineffective estrogen suppression (SES) (with E2 > 2.72 pg/mL, or any vaginal bleeding > 3 months after triptorelin start or pregnancy) such as: age, evidence of menses at entry, BMI, chemotherapy (yes/no), and, type of chemotherapy received
Time Frame: Four years after randomization
Population: All patients from the Intent to treat (ITT) population assigned to exemestane +triptorelin (N=83) according to suboptimal estrogen suppression (SES) with E2 > 2.72 pg/mL (suboptimal threshold) or any vaginal bleeding > 3 mos after triptorelin start or pregnancy
Measure: Count of Participants; unit: Participants
Groups:
- Triptorelin Plus Exemestane With Suboptimal Estrogen Suppression (E2>2.72 pg/mL); Triptorelin Plus Exemestane Without Suboptimal Estrogen Suppression (E2>2.72 pg/mL): Determination of estrogen levels in blood samples from patients being treated with triptorelin plus exemestane for 5 years.
Arm/Group | Triptorelin Plus Exemestane With Suboptimal Estrogen Suppression (E2>2.72 pg/mL) | Triptorelin Plus Exemestane Without Suboptimal Estrogen Suppression (E2>2.72 pg/mL)
Number analyzed (Participants) | 21 | 62
Participants
  Age at randomization (years), <35 | 3 | 5
  Age at randomization (years), >=35 | 18 | 57
  Menstrual status, normal | 13 | 24
  Menstrual status, irregular | 3 | 11
  Menstrual status, persistent amenorrhea | 5 | 27
  BMI (kg/m2), normal (<25) | 9 | 36
  BMI (kg/m2), over weight (25-<30) | 8 | 16
  BMI (kg/m2), obese (>=30) | 3 | 9
  Prior chemo, no | 12 | 25
  Prior chemo, yes | 9 | 37
  Prior chemo regimen, no chemo | 12 | 25
  Prior chemo regimen, anthracycline-based | 3 | 7
  Prior chemo regimen, taxane-based | 0 | 2
  Prior chemo regimen, anthracycline+taxane | 6 | 28

5. Secondary Outcome: Baseline Estrogen Levels (E2, E1, E1S) With Suboptimal Estrogen Suppression (SES) in the Exemestane + Triptorelin Arm
Description: The secondary analysis explored baseline estrogen levels (E2, E1, E1S) with suboptimal estrogen suppression (SES) where estrogen (E2) > 2.72 pg/mL in the exemestane + triptorelin arm.
Time Frame: Baseline
Population: as for outcome 4
Measure: Median (Inter-Quartile Range); unit: pg/mL
Groups:
- Triptorelin Plus Exemestane With Suboptimal Estrogen Suppression (SES) With E2>2.72 pg/mL; Triptorelin Plus Exemestane Without Suboptimal Estrogen Suppression (SES) With E2>2.72 pg/mL: Determination of estrogen levels in blood samples from patients being treated with triptorelin plus exemestane for 5 years.
Arm/Group | Triptorelin Plus Exemestane With Suboptimal Estrogen Suppression (SES) With E2>2.72 pg/mL | Triptorelin Plus Exemestane Without Suboptimal Estrogen Suppression (SES) With E2>2.72 pg/mL
Number analyzed (Participants) | 21 | 62
pg/mL
  Baseline estradiol (E2) | 80 [60 to 121] | 39 [6 to 83]
  Baseline estrone (E1) | 50 [26 to 59] | 41 [23 to 71]
  Baseline estrone sulphate (E1S) | 928 [572 to 1168] | 715 [302 to 1330]

6. Secondary Outcome: Baseline Endocrine Function Levels (FSH, LH) With Suboptimal Estrogen Suppression (SES) in the Exemestane + Triptorelin Arm
Description: The secondary analysis explored endocrine functions (FSH, LH) with suboptimal estrogen suppression (SES) where estrogen (E2) > 2.72 pg/mL in the exemestane + triptorelin arm.
Time Frame: Baseline
Population: as for outcome 4
Measure: Median (Inter-Quartile Range); unit: IU/L
Arm/Group | Triptorelin Plus Exemestane With Suboptimal Estrogen Suppression (SES) With E2>2.72 pg/mL | Triptorelin Plus Exemestane Without Suboptimal Estrogen Suppression (SES) With E2>2.72 pg/mL
Number analyzed (Participants) | 21 | 62
IU/L
  Baseline follicle-stimulating hormone (FSH) | 6 [5 to 8] | 32 [10 to 58]
  Baseline luteinizing hormone (LH) | 6 [4 to 8] | 21 [7 to 32]

7. Secondary Outcome: Endocrine Functions (FSH and LH) Status According to Treatment Assignments
Description: Endocrine function (FSH, LH) status according to treatment assignments at 12 months using 12 month data alone or 12 month data plus earlier data (when 12 month not available)
Time Frame: Less than 12 months, at 12 months
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: IU/L
Arm/Group | Triptorelin Plus Tamoxifen | Triptorelin Plus Exemestane
Number analyzed (Participants) | 26 | 83
IU/L
  Follicle-stimulating hormone (FSH) at 12 months | 2.0 [1.5 to 2.6] | 7.0 [5.2 to 8.8]
  Follicle-stimulating hormone (FSH) at <=12 months | 2.2 [1.6 to 3.1] | 6.5 [4.8 to 8.7]
  Luteinizing hormone (LH) at 12 months | 0.2 [0.1 to 0.4] | 0.1 [0.1 to 0.1]
  Luteinizing hormone (LH) at <=12 months | 0.2 [0.1 to 0.4] | 0.1 [0.1 to 0.2]

ADVERSE EVENTS:
Time Frame: Four years after randomization.
Description: Adverse event data were not collected for the substudy population but were for the main study.
Arm/Group | Triptorelin Plus Tamoxifen | Triptorelin Plus Exemestane
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No